CLINICAL TRIAL: NCT03760497
Title: Comparison of Three Restorative Protocols in Teeth With Molar-Incisor Hipomineralization (MIH): a Randomized Controlled Clinical Study
Brief Title: Three Restorative Protocols in MIH: a Randomized Controlled Clinical Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Vicioni-Marques, F, Comparison of Three Restorative Protocols in Teeth With Molar-Incisor Hipomineralization (MIH): a Randomized Controlled Clinical Study, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MIHFORPUSP
Record Dates: First submitted 2018-11-27; First posted 2018-11-30 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Molar Incisor Hypomineralization
Keywords: Lasers; Hipomineralization of dental enamel; Preventive dentistry; Glass ionomer cement
MeSH Terms: conditions — Molar Hypomineralization | interventions — Dental Atraumatic Restorative Treatment

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- CIV Group (Experimental): Temporary Restoration with Glass Ionomer (Equia Forte® - GC Corporation, Tokyo, Japan) for 30 days + Restoration in Composite Resin (Filtek® Resin Z350 XT - 3M Corporate Headquarters, St. Paul, USA).
  Interventions: Procedure: Restorative treatment
- Composite Resin Group (Experimental): Restoration with Composite Resin (Filtek® Resin Z350 XT - 3M Corporate Headquarters, St. Paul, United States).
  Interventions: Procedure: Restorative treatment
- Composite Resin Group + Laser (Experimental): Composite Resin Restoration (Filtek® Resin Z350 XT - 3M Corporate Headquarters, St. Paul, USA) + Application of Diode Laser.
  Interventions: Procedure: Restorative treatment

INTERVENTIONS:
Procedure: Restorative treatment — For all groups, first the patients will be submitted to the anesthetic technique indicated with Lidocaine + Epinephrine 1: 100,000 (New DFL, Rio de Janeiro, Brazil), followed by absolute isolation with rubber sheet and metal clamp; then prophylaxis of the selected tooth will be performed with Robson's brush and pumice stone and water, surface washing and drying with cotton balls, removal of carious tissue or affected enamel without dentin support with sharp curettes or low-speed spherical drills. Subsequently, each group will follow the treatment protocols suggested by the manufacturer of restorative materials.

SUMMARY:
Molar-Incisive Hipomineralization (MIH) is defined as a qualitative change in tooth enamel of systemic origin, which affects one or more permanent first molars, and may or may not involve permanent incisors. MIH has several clinical repercussions, such as presence of hypersensitivity, difficulty in local anesthesia, reduction of restorations longevity, among others, making it difficult to perform dental treatment. Therefore, the present study will evaluate, through a randomized controlled clinical study, three restorative protocols for the treatment of severe MIH (with post eruptive enamel fracture and dentin exposure). The following groups will be evaluated: direct restoration with composite resin; restoration with composite resin with diode laser application and temporary restoration with glass ionomer cement followed by restoration with composite resin). The restorations will be evaluated after 1 week, 1, 6, 12, 18 and 24 months. The main outcome will be evaluation of restoration longevity, presence of caries lesion and wear of the restoration surface. Other outcomes such as patient satisfaction with treatment, patient discomfort, anxiety, assessment of dentin sensitivity and impact on participants' quality of life, as well as the duration and cost of treatment, as well as their cost-effectiveness ratio will also be evaluated . Multilevel statistical analyzes will be performed to verify the effectiveness of diode laser treatment compared to sealing, in addition to possible factors associated with this efficacy.

ELIGIBILITY:
Inclusion Criteria:

- At least one permanent first molar with occlusal surface with severe MIH grade (with post eruptive enamel fracture and dentin exposure), it may not be reported hypersensitivity in the selected tooth.

Exclusion Criteria:

-

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2021-12 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Longevity of restorations | 24 months.
  The main purpose will be the longevity of the desserts in elaborate compounds, according to the three protocols.
  Images should be analyzed and scanned. Radiographic examination and digital radiography. After 6, 12 and 24 months.
Treatment satisfaction as assessed by VAS scale (Index 0 to 10) | After 1 week of treatment, 1, 12 and 24 months.
  After 1 week of treatment, 1, 12 and 24 months, the caregiver will be asked to respond about the satisfaction regarding the care (treatment and returns) received. He should classify his satisfaction using the VAS scale with indexes from 0 to 10, with 0 being the worst treatment evaluation and 10 being the best.
Discomfort referred by the children assessed by Wong-Baker Facial Scale (Very smiling to very sad) | On treatment day
  In order to assess the discomfort reported by the children in relation to the type of treatment received, the same timekeeping operator will apply the Wong-Baker Facial Scale to the patient, which is composed of six figures with equidistant faces. that the first one is very smiling and the expressions are changing, until the last one is very sad.
Quality of life assessed by Child Perceptions Questionnaire 8-10 (CPQ8-10) (Assessed by questions) | On treatment day
  To assess the impact of MIH on children's quality of life, the Child Perceptions Questionnaire 8-10 (CPQ8-10), specially developed for children aged 8-10 years and validated in the Portuguese language. This scale was assessed through questions and answers to a children's quality of life.
Anxiety Assessment | On treatment day
  For the assessment of anxiety in the study children, the Children's Fear Survey Schedule-Dental Subscale will be used

SECONDARY OUTCOMES:
Socioeconomic questionnaire | On treatment day
  Information obtained through a socioeconomic questionnaire and questions related to the individual characteristics of the child, such as, for example, fluoride exposure variables, oral hygiene practices and eating habits.
Evaluation of the caries experience | On treatment day
  Evaluation of the caries experience by the ceo-d / CPO-D indices
Presence of biofilm visible | On treatment day
  Presence of biofilm visible through the Simplified Oral Hygiene Index in which six surfaces will be used to represent the entire mouth: the vestibular of the first right and left first molars, the lingual of the first right and left first molars, and the vestibular surface of the upper central incisor right and bottom left
Evaluation of the visible biofilm accumulated on the occlusal surface | On treatment day
  First the presence of dental biofilm will be evaluated visually, according to the following index: 0: absence of visible biofilm; 1: visible but difficult to identify biofilm - best verified after drying; 2: Visible and easily identifiable biofilm - even without drying
Evaluation of the presence of visible biofilm on the buccal surfaces of the molars to be evaluated | On treatment day
  0: absence of visible biofilm, 1: biofilm not visible, but removed from the gingival sulcus with the periodontal probe; 2: visible biofilm after drying; 3: abundant biofilm, visible even without drying.
Assessment of eruption degree | On treatment day
  The degree of eruption will be assessed according to the following criteria (5): A: not erupted or less than 1/3 of the erupted occlusal surface or part of the crown of the visible incisor; B: totally erupted or at least 1/3, but less than the total occlusal surface erupted and / or less than the total crown length of the visible incisor.
Evaluation of lesion extension | On treatment day
  The extent of lesion will be evaluated according to the following criterion (5): I: less than one third of the affected tooth, II: at least 1/3 of the affected tooth, but less than 2/3, III : at least 2/3 of the affected tooth.
Cost of procedures | On treatment day
  To calculate the direct costs of the procedures, the time spent in each consultation (initials and reevaluations) will be taken into account. The time will be timed and recorded in a specific clinical record. For the calculation of direct costs, the prices of consumer and permanent materials (specifications and quantity) used in each procedure, electricity and the professional fee will be considered. These values will be inferences of the market value obtained by average of different places that market the products in question, being updated during the time of the study. In addition, the cost of equipment depreciation and electricity will be calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- School of Dentistry of Ribeirao Preto, Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided